CLINICAL TRIAL: NCT05819021
Title: An Open Label Optimization Study to Assess the Effectiveness of the SAINT® Neuromodulation System (NMS) to Treat Major Depressive Disorder
Brief Title: Open Label Optimization Study
Acronym: OLO
Status: Active, not recruiting | Type: Observational
Sponsor: Magnus Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0107
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SAINT® Stimulation: All participants will receive 10 treatments per day for 5 days (M-F) of SAINT® stimulation therapy.
  Interventions: Device: SAINT® Neuromodulation System (NMS)

INTERVENTIONS:
Device: SAINT® Neuromodulation System (NMS) — The SAINT® NMS utilizes a type of accelerated iTBS delivered to a personalized treatment target derived from a functional MRI scan. SAINT® was designed to optimize the individual patient response to treatment. This novel approach to TMS is accomplished by focusing on three critical aspects of the treatment that drive effect. These aspects are personalized stimulation target, total course dose of stimulation, and neurophysiologically relevant stimulation pattern.
  Other Names: TMS

SUMMARY:
The goal of this observational study is to demonstrate effectiveness in the treatment of Major Depressive Disorder

The primary objective is to assess the effectiveness in the treatment of Major Depressive Disorder using the CGI-I at the end of the treatment

Participants will receive 10 treatments per day for 5 days (M-F) of SAINT®

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label study.

Up to 1000 adult subjects, in a major depressive episode, who have failed to receive satisfactory improvement from a prior antidepressant medication in the current episode, are eligible to participate in this study if they are deemed to be appropriate candidates for TMS.

Overall study duration is expected to be approximately 4 years. The study duration per subject is anticipated to be approximately 1 year.

Hypothesis: The SAINT® Neuromodulation System will demonstrate effectiveness in the treatment of MDD as measured by CGI-I at the end of the treatment (cessation of stimulation).

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females, 18 and older, who have failed to receive satisfactory improvement from prior antidepressant medication in the current episode.
2. Confirmed primary clinical diagnosis of major depressive disorder (MDD) without psychotic features consistent with DSM-V criteria.
3. No medical conditions that would preclude the safe use of TMS.
4. Primary psychiatrist has determined TMS to be an appropriate clinical option.
5. Able to provide consent and comply with all study requirements.
6. Negative pregnancy test at the intended time of SAINT™ 5-day acute course treatment and agreement to use effective birth control during SAINT® acute therapy.

Exclusion Criteria:

1. Have any contraindication to TMS (section 2 User Manual).
2. Have any contraindication to receiving an MRI
3. Participants with an abnormal brain MRI as determined by PI, study physician or designee.
4. Deemed by the PI, study physician or designee to be a high risk of suicide or has made a suicide attempt within the last 6 months.
5. Treatment dose with cortical depth adjustment is greater than 120% motor threshold and cannot be completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who fulfill all the inclusion criteria and none of the exclusion criteria will be enrolled into the study. Each participant will read and sign the IRB approved informed consent form prior to any screening or study procedures being performed. This open-label study involves an evaluation of the safety and effectiveness of an acute course of the SAINT® NMS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Mean Clinical Global Impression Improvement Scale (CGI-I) score at the end of treatment (Day 5 SAINT® therapy) | End of Stimulation Day 5
  Clinical Global Impression-Improvement (CGI-I) score is based on a scale from zero (0) - Not Assessed to seven (7) Very Much Worse with lower scores showing improvement and higher scores showing little or no improvement.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) score change from baseline to cessation of stimulation in comparison with bioimaging assessments MADRS score change from baseline to cessation of stimulation in comparison with bioimaging assessments | Baseline to End Stimulation Day 5
  The rating is based on a clinical interview. Questions are asked using scales from zero (0) to six (6) with lower scores showing a better outcome and higher scores showing a worse outcome
Cambridge Brain Science Tools assessment score change in comparison with change in MADRS scores from baseline to cessation of stimulation | Baseline to End of Stimulation Day 5
  Assess aspects of cognition including reasoning, memory, attention and verbal ability on an online platform. Scores are automatically calculated on a scale from zero (0) to one hundred (100) and zero (0) to negative one hundred (-100) with positive numbers being associated with "Best" and negative numbers being associated with "Worst"
To test the durability of the antidepressant effect by assessing the Clinical Global Impression Severity Scale (CGI-S) after cessation of stimulation | 3, 6, 9, 12 month follow up visit
  The Clinical Global Impression-Severity (CGI-S) is a brief clinician assessment that rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Score is based on a scale from zero (0) - Not Assessed to seven (7) Very Much Worse with lower scores showing improvement and higher scores showing little or no improvement.

OTHER OUTCOMES:
Safety - Adverse Event Reporting assessment for causality and severity | Consent through 12 month follow up visit
  Any untoward medical occurrence in a participant treated with an investigational device, without regard to the possibility of a causal relationship with this treatment. Adverse events will be recorded and followed through all follow-up visits

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - BrainHealth Solutions, Costa Mesa, California
  - LA TMS, Los Angeles, California
  - Integral TMS, Sunnyvale, California
  - Acacia Research Center, Sunnyvale, California
  - Boston Precision Neurotherapeutics, Natick, Massachusetts
  - Fermata, Brooklyn, New York
  - Seattle Neuropsychiatric Treatment Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided